CLINICAL TRIAL: NCT06113666
Title: Digital Cognitive Behavior Therapy for Insomnia Compared With Digital Patient Education About Insomnia in People With Multiple Sclerosis in Norway
Brief Title: A Digital Therapeutic to Improve Insomnia in Multiple Sclerosis: A Randomized Controlled Trial.
Acronym: NorseMS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: St. Olavs Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 623308
Record Dates: First submitted 2023-10-27; First posted 2023-11-02 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Multiple Sclerosis; Insomnia
Keywords: Cognitive Behavioral Therapy for Insomnia; Fatigue; Cognitive performance
MeSH Terms: conditions — Multiple Sclerosis; Sleep Initiation and Maintenance Disorders; Fatigue

STUDY DESIGN:
Masking Description: The participants are in theory blinded to which group they are allocated to. However, it is not possible to blind completely as it is easy for the patients to see if they are receiving active, interactive treatment or are allocated into the control group with patient education.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Digital cognitive behavioral therapy for insomnia (Experimental): Behavioral: digital cognitive behavioral therapy (dCBT-I)
  Interventions: Behavioral: Digital Cognitive Behavioral Therapy for Insomnia (dCBT-I)
- Patient Education about insomnia (Active Comparator): Behavioral: Digital patient education about insomnia (PE)
  Interventions: Behavioral: Digital patient education about insomnia (PE)

INTERVENTIONS:
Behavioral: Digital Cognitive Behavioral Therapy for Insomnia (dCBT-I) — dCBT-I during 9 weeks. Multicomponent intervention that includes the following: psychoeducation about sleep, sleep hygiene, sleep restriction therapy, stimulus control and challenging beliefs and perception about sleep. The digital CBT-I that will be utilized in this study is named Sleep Healthy Using The internet (SHUTi). The intervention is fully automated with no contact with health care personnel, it is interactive and adapts to input from the users. It comprises of the same elements included in face-to-face CBT-I, but the user gains access to a new educational, behavioral or cognitive module each week only after completion of digital sleep diaries. dCBT-I can be accessed on computers or hand-held devices
  Other Names: Sleep Healthy Using The Internet (SHUTi)
  Arms: Digital cognitive behavioral therapy for insomnia
Behavioral: Digital patient education about insomnia (PE) — Control condition PE during 9 weeks. A digital patient education program that can be accessed on computers or hand-held devices. The information overlaps with that included in the dCBT-I intervention but it does not include any of the interactive features of the dCBT-I intervention and all the information is available from the moment the PE site is opened.
  Arms: Patient Education about insomnia

SUMMARY:
The goal of this randomized controlled trial is to test the effectiveness of digital cognitive behavioral therapy for insomnia (dCBT-I) compared with digital patient education about insomnia for people with Multiple Sclerosis (MS). The main questions it aims to answer are whether dCBT-I is effective in reducing insomnia severity in people with MS, whether dCBT-I is effective in reducing daytime fatigue, psychological distress, cognitive problems, medication use (hypnotic, sedative/anxiolytic and antidepressant), resource utilization and if these changes are mediated by improvements in insomnia severity and whether dCBT-I is feasible for people with MS

DETAILED DESCRIPTION:
Insomnia is prevalent among individuals with Multiple Sclerosis (MS). Improving sleep is an important therapeutic goal, but there is currently a lack of effective treatment options. Cognitive Behavioral Therapy for Insomnia (CBT-I) has been widely studied in other patient groups and is currently recommended as first- line treatment for chronic insomnia.

Overall, the availability of CBT-I has been limited, as the number of patients in need of treatment far exceeds the number of available therapists. Therefore, fully automated digital adaptations of CBT-I (dCBT-I) have been developed that contain both screening and intervention. Whether this treatment is effective for a clinical sample of patients diagnosed with MS, or if improved sleep can lead to improved daytime functioning in MS, is however, currently unknown.

This is a novel approach to a digital treatment of a common disorder in MS, and that may result in improved implementation of a low-threshold intervention.

Update August 28th, 2024

We aim to increase the target sample size from 260 to 550 to increase the statistical power to detect differences between the intervention group and control group on the secondary outcomes, e.g., fatigue, cognitive functioning, mental health, and movement measures measured with actigraphy. Few treatment options have shown effects on these outcomes for people with MS but are a significant problem for this patient group. Small effects from this trial may have substantial scientific and clinical value and are important to test with adequate statistical power.

Based on previous RCTs investigating the effectiveness of dCBT-I we aim to have a sample size large enough to detect small to moderate effects (Cohen's d = 0.3 til 0.5) on the secondary outcome measures fatigue, cognitive function, mental health and movement measures measured with actigraphy. As the planned RCT involves limited contact between researchers and participants, we have predicted that the study dropout rate will likely reach about 50%. Therefore, we aim to recruit 550 participants, to enable us to retain 275 participants (137 in each treatment arm) at the end of the RCT. For a two-sample t-test with alpha=0.05, this sample size gives a power of 90% of detecting a difference of Cohen's d = 0.40.

ELIGIBILITY:
Inclusion Criteria:

1. Having an established diagnosis of Multiple Sclerosis (MS) and being included in the Norwegian MS registry
2. Being 18 years or older
3. Scoring at least 12 points on the Insomnia Severity Index
4. Willing and able to provide written informed consent

Exclusion Criteria:

1. Self-reported symptoms of sleep apnea: Positive endorsement of a screening question for sleep apnoea (the item asks if they 'usually or everyday snore and stop breathing and have difficulties staying awake during the day')
2. Self-reported surgery for heart disease the last two months
3. Currently in an attack phase of MS and/or on treatment with steroids,
4. Self-reported night shifts in their work schedule,
5. Inadequate opportunity to sleep or living in circumstances that prevent modification of sleep pattern (e.g. having an infant residing at home),
6. Pregnant in the last two trimesters
7. Unable to get into bed or out of bed without human assistance.
8. Concomitant psychological treatment for sleep problems

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 550 (Estimated)
Dates: Start 2023-11-16 (Actual); Primary Completion 2025-10-30 (Estimated); Study Completion 2029-10-30 (Estimated)

PRIMARY OUTCOMES:
Between-group difference in insomnia severity at week 9 after randomization | 9 weeks after randomization
  Assessed with the Insomnia Severity Index (ISI), a 7-item questionnaire for the severity of insomnia symptoms the last 14 days. Each item is rated on a 0 to 4 rating scale with higher scores indicating more severe symptoms. The ISI has good psychometric properties and is validated for online use. Range is 0-28 with higher values represent higher levels of insomnia symptom severity.

SECONDARY OUTCOMES:
Between-group difference in insomnia severity at week 33 after randomization | 33 weeks after randomization
  While between-group difference on the ISI on week 9 is our primary endpoint, we will also assess between group differences on the ISI at week 33 (six months after post-assessment) and week 61 (one year after post assessment). Assessed with the Insomnia Severity Index (ISI), a 7-item questionnaire for the severity of insomnia symptoms the last 14 days. Each item is rated on a 0 to 4 rating scale with higher scores indicating more severe symptoms. The ISI has good psychometric properties and is validated for online use. Range is 0-28 with higher values represent higher levels of insomnia symptom severity.
Between-group difference in insomnia severity at week 61 after randomization | 61 weeks after randomization
  While between-group difference on the ISI on week 9 is our primary endpoint, we will also assess between group differences on the ISI at week 33 (six months after post-assessment) and week 61 (one year after post assessment). Assessed with the Insomnia Severity Index (ISI), a 7-item questionnaire for the severity of insomnia symptoms the last 14 days. Each item is rated on a 0 to 4 rating scale with higher scores indicating more severe symptoms. The ISI has good psychometric properties and is validated for online use. Range is 0-28 with higher values represent higher levels of insomnia symptom severity.
Prospective daily sleep-wake pattern at week 9 after randomization | 9 weeks after randomization
  Assessed with the Consensus Sleep Dairy (sleep-onset latency [SOL]; wake-time after sleep onset [WASO]; sleep efficiency [SE]; total sleep time [TST]; sleep quality [SQ]), which will be completed by the participant at baseline and each follow-up point for at least 10 out of 14 consecutive days.
Prospective daily sleep-wake pattern at week 33 after randomization | 33 weeks after randomization
  Assessed with the Consensus Sleep Dairy (sleep-onset latency [SOL]; wake-time after sleep onset [WASO]; sleep efficiency [SE]; total sleep time [TST]; sleep quality [SQ]), which will be completed by the participant at baseline and each follow-up point for at least 10 out of 14 consecutive days.
Prospective daily sleep-wake pattern at week 61 after randomization | 61 weeks after randomization
  Assessed with the Consensus Sleep Dairy (sleep-onset latency [SOL]; wake-time after sleep onset [WASO]; sleep efficiency [SE]; total sleep time [TST]; sleep quality [SQ]), which will be completed by the participant at baseline and each follow-up point for at least 10 out of 14 consecutive days.
Self-reported mental health status at baseline | Baseline
  Assessed with the Outcome Questionnaire - 45.2 (OQ-45.2), a 45 item self-report scale for mental health status, specifically designed for patient progress throughout therapy. It has excellent internal consistency and is highly correlated with well-known outcomes such as the Symptom Checklist 90R, Beck Depression Inventory, The State Trait Inventory, The inventory of interpersonal problems, The Social Adjustment Scale, and the SF-36.34 The scale is scored on a scale of 0 (=never) to 5 (=almost always) giving a range of 0 to 180, with higher scores indicating higher levels of psychopathology. The OQ-45.2 has three validated subscales: symptom distress, interpersonal relations, and social role functioning (perceived level of difficulties in the workplace, school or home duties). Results will be reported for the sum score, and for the three subscales. The OQ-45.2 has an established clinical cut-off value and reliable change index
Self-reported mental health status at week 9 after randomization | 9 weeks after randomization
  Assessed with the Outcome Questionnaire - 45.2 (OQ-45.2), a 45 item self-report scale for mental health status, specifically designed for patient progress throughout therapy. It has excellent internal consistency and is highly correlated with well-known outcomes such as the Symptom Checklist 90R, Beck Depression Inventory, The State Trait Inventory, The inventory of interpersonal problems, The Social Adjustment Scale, and the SF-36.34 The scale is scored on a scale of 0 (=never) to 5 (=almost always) giving a range of 0 to 180, with higher scores indicating higher levels of psychopathology. The OQ-45.2 has three validated subscales: symptom distress, interpersonal relations, and social role functioning (perceived level of difficulties in the workplace, school or home duties). Results will be reported for the sum score, and for the three subscales. The OQ-45.2 has an established clinical cut-off value and reliable change index
Self-reported mental health status at week 33 after randomization | 33 weeks after randomization
  Assessed with the Outcome Questionnaire - 45.2 (OQ-45.2), a 45 item self-report scale for mental health status, specifically designed for patient progress throughout therapy. It has excellent internal consistency and is highly correlated with well-known outcomes such as the Symptom Checklist 90R, Beck Depression Inventory, The State Trait Inventory, The inventory of interpersonal problems, The Social Adjustment Scale, and the SF-36.34 The scale is scored on a scale of 0 (=never) to 5 (=almost always) giving a range of 0 to 180, with higher scores indicating higher levels of psychopathology. The OQ-45.2 has three validated subscales: symptom distress, interpersonal relations, and social role functioning (perceived level of difficulties in the workplace, school or home duties). Results will be reported for the sum score, and for the three subscales. The OQ-45.2 has an established clinical cut-off value and reliable change index
Self-reported mental health status at week 61 after randomization | 61 weeks after randomization
  Assessed with the Outcome Questionnaire - 45.2 (OQ-45.2), a 45 item self-report scale for mental health status, specifically designed for patient progress throughout therapy. It has excellent internal consistency and is highly correlated with well-known outcomes such as the Symptom Checklist 90R, Beck Depression Inventory, The State Trait Inventory, The inventory of interpersonal problems, The Social Adjustment Scale, and the SF-36.34 The scale is scored on a scale of 0 (=never) to 5 (=almost always) giving a range of 0 to 180, with higher scores indicating higher levels of psychopathology. The OQ-45.2 has three validated subscales: symptom distress, interpersonal relations, and social role functioning (perceived level of difficulties in the workplace, school or home duties). Results will be reported for the sum score, and for the three subscales. The OQ-45.2 has an established clinical cut-off value and reliable change index
Anxiety/depression at baseline | Baseline
  Assessed with the Hospital Anxiety and Depression Scale (HADS), a 14-item questionnaire for non-vegetative symptoms of anxiety and depression on a 0 to 3 likert scale. The sum score can be used as a measure of general psychological distress and is widely used in the community, general practice and psychiatric settings. It has a range of 0 to 42 points with higher scores indicating higher levels of psychological distress.
Anxiety/depression at week 9 after randomization | 9 weeks after randomization
  Assessed with the Hospital Anxiety and Depression Scale (HADS), a 14-item questionnaire for non-vegetative symptoms of anxiety and depression on a 0 to 3 likert scale. The sum score can be used as a measure of general psychological distress and is widely used in the community, general practice and psychiatric settings. It has a range of 0 to 42 points with higher scores indicating higher levels of psychological distress.
Anxiety/depression at week 33 after randomization | 33 weeks after randomization
  Assessed with the Hospital Anxiety and Depression Scale (HADS), a 14-item questionnaire for non-vegetative symptoms of anxiety and depression on a 0 to 3 likert scale. The sum score can be used as a measure of general psychological distress and is widely used in the community, general practice and psychiatric settings. It has a range of 0 to 42 points with higher scores indicating higher levels of psychological distress.
Anxiety/depression at week 61 after randomization | 61 weeks after randomization
  Assessed with the Hospital Anxiety and Depression Scale (HADS), a 14-item questionnaire for non-vegetative symptoms of anxiety and depression on a 0 to 3 likert scale. The sum score can be used as a measure of general psychological distress and is widely used in the community, general practice and psychiatric settings. It has a range of 0 to 42 points with higher scores indicating higher levels of psychological distress.
Fatigue at baseline | Baseline
  Assessed with the Chalder Fatigue Questionnaire (CFQ), a 11-item questionnaire for daytime physical and psychological fatigue on a 0 to 3 likert scale (0=less than usual, 3=much more than usual). The scale has a range of 0 to 33 with higher scores indicating higher levels of fatigue. Two additional items assess duration of fatigue (0=less than a week, 4=six months or more) and how much of the time the individual experience fatigue (0=25% of the time, 3=all the time)
Fatigue at week 9 after randomization | 9 weeks after randomization
  Assessed with the Chalder Fatigue Questionnaire (CFQ), a 11-item questionnaire for daytime physical and psychological fatigue on a 0 to 3 likert scale (0=less than usual, 3=much more than usual). The scale has a range of 0 to 33 with higher scores indicating higher levels of fatigue. Two additional items assess duration of fatigue (0=less than a week, 4=six months or more) and how much of the time the individual experience fatigue (0=25% of the time, 3=all the time)
Fatigue at week 33 after randomization | 33 weeks after randomization
  Assessed with the Chalder Fatigue Questionnaire (CFQ), a 11-item questionnaire for daytime physical and psychological fatigue on a 0 to 3 likert scale (0=less than usual, 3=much more than usual). The scale has a range of 0 to 33 with higher scores indicating higher levels of fatigue. Two additional items assess duration of fatigue (0=less than a week, 4=six months or more) and how much of the time the individual experience fatigue (0=25% of the time, 3=all the time)
Fatigue at week 61 after randomization | 61 weeks after randomization
  Assessed with the Chalder Fatigue Questionnaire (CFQ), a 11-item questionnaire for daytime physical and psychological fatigue on a 0 to 3 likert scale (0=less than usual, 3=much more than usual). The scale has a range of 0 to 33 with higher scores indicating higher levels of fatigue. Two additional items assess duration of fatigue (0=less than a week, 4=six months or more) and how much of the time the individual experience fatigue (0=25% of the time, 3=all the time)
Fatigue severity at baseline | Baseline
  Assessed with the Fatigue Severity Scale (FSS), a 9-item questionnaire with statements about physical, social and cognitive effects of fatigue on a 1 to 7 likert scale (1=strongly disagree, 7=strongly agree). Higher total scores indicate higher levels of fatigue.
Fatigue severity at week 9 after randomization | 9 weeks after randomization
  Assessed with the Fatigue Severity Scale (FSS), a 9-item questionnaire with statements about physical, social and cognitive effects of fatigue on a 1 to 7 likert scale (1=strongly disagree, 7=strongly agree). Higher total scores indicate higher levels of fatigue.
Fatigue severity at week 33 after randomization | 33 weeks after randomization
  Assessed with the Fatigue Severity Scale (FSS), a 9-item questionnaire with statements about physical, social and cognitive effects of fatigue on a 1 to 7 likert scale (1=strongly disagree, 7=strongly agree). Higher total scores indicate higher levels of fatigue.
Fatigue severity at week 61 after randomization | 61 weeks after randomization
  Assessed with the Fatigue Severity Scale (FSS), a 9-item questionnaire with statements about physical, social and cognitive effects of fatigue on a 1 to 7 likert scale (1=strongly disagree, 7=strongly agree). Higher total scores indicate higher levels of fatigue.
Cognitive test performance at baseline | Baseline
  Assessed with the home-based cognitive test battery Memoro. At baseline the test battery includes subtests for assessing reaction time, spatial memory, working memory, processing speed, attention and abstract reasoning.
Cognitive test performance at week 9 after randomization | 9 weeks after randomization
  Assessed with the home-based cognitive test battery Memoro. At follow-up the test battery includes the subtests Coding (The Symbol Digit Modalities Test) assessing processing speed and a continuous performance test assessing attention and cognitive control function. Cognitive performance will be assessed with reaction time, number of errors and performance variability (standard deviations of hit reaction times).
Cognitive test performance at week 33 after randomization | 33 weeks after randomization
  Assessed with the home-based cognitive test battery Memoro. At follow-up the test battery includes the subtests Coding (The Symbol Digit Modalities Test) assessing processing speed and a continuous performance test assessing attention and cognitive control function. Cognitive performance will be assessed with reaction time, number of errors and performance variability (standard deviations of hit reaction times).
Cognitive test performance at week 61 after randomization | 61 weeks after randomization
  Assessed with the home-based cognitive test battery Memoro. At follow-up the test battery includes the subtests Coding (The Symbol Digit Modalities Test) assessing processing speed and a continuous performance test assessing attention and cognitive control function. Cognitive performance will be assessed with reaction time, number of errors and performance variability (standard deviations of hit reaction times).
Continuous recordings of daytime activity and sleep from baseline to 9 weeks after randomization | From baseline to 9 weeks after randomization.
  Sleep and daytime activity will be recorded using actigraphy (GENEactiv Original, Activinsights Ltd, Kimbolton, United Kingdom). This will primarily allow collection of data to assess details of sleep-wake cycles as well as adherence to the intervention. It will also allow assessment of any intervention-related changes in daytime activity patterns and novel use of mathematical modelling.
Use of health care services at baseline | Baseline
  Number of appointments at mental health care clinics, type and timing of treatment and admissions, and date of the first appointment for each patient during the study period from the Norwegian Patient Registry
Use of health care services at 61 weeks after randomization | 61 weeks after randomization
  Number of appointments at mental health care clinics, type and timing of treatment and admissions, and date of the first appointment for each patient during the study period from the Norwegian Patient Registry
Use of health care services at 5 years after randomization | 5 years after randomization
  Number of appointments at mental health care clinics, type and timing of treatment and admissions, and date of the first appointment for each patient during the study period from the Norwegian Patient Registry
Medication use at baseline | Baseline
  Dose, timing, and type of prescribed hypnotic, sedative/anxiolytic, antidepressant and other psychotropic medications and medications used in treatment of MS (According to the WHO Anatomical Therapeutic Chemical Classification System) and changes recorded during the RCT (data from the Norwegian Prescription Database
Medication use at 61 weeks after randomization | 61 weeks after randomization
  Dose, timing, and type of prescribed hypnotic, sedative/anxiolytic, antidepressant and other psychotropic medications and medications used in treatment of MS (According to the WHO Anatomical Therapeutic Chemical Classification System) and changes recorded during the RCT (data from the Norwegian Prescription Database
Medication use at 5 years after randomization | 5 years after randomization
  Dose, timing, and type of prescribed hypnotic, sedative/anxiolytic, antidepressant and other psychotropic medications and medications used in treatment of MS (According to the WHO Anatomical Therapeutic Chemical Classification System) and changes recorded during the RCT (data from the Norwegian Prescription Database
Costs of treatment offered by the public services at baseline | Baseline
  Data from the database named 'Kontroll og Utbetaling av Helserefusjon'
Costs of treatment offered by the public services 61 weeks after randomization | 61 weeks after randomization
  Data from the database named 'Kontroll og Utbetaling av Helserefusjon'
Costs of treatment offered by the public services 5 years after randomization | 5 years after randomization
  Data from the database named 'Kontroll og Utbetaling av Helserefusjon'
Sick leave or in receipt of disability benefits at baseline | Baseline
  Data from the administrative database called Forløpsdatabasen
Sick leave or in receipt of disability benefits 61 weeks after randomization | 61 weeks after randomization
  Data from the administrative database called Forløpsdatabasen
Sick leave or in receipt of disability benefits 5 years after randomization | 5 years after randomization
  Data from the administrative database called Forløpsdatabasen
Information about the MS disease at baseline | Baseline
  Disability status assessed with the Extended Disability Status Scale from the Norwegian MS registry, information about previous and current treatment for MS, previous attack phases, first diagnosis of MS from the Norwegian MS registry.
Information about the MS disease at week 61 after randomization | 61 weeks after randomization
  Disability status assessed with the Extended Disability Status Scale from the Norwegian MS registry, information about previous and current treatment for MS, previous attack phases, first diagnosis of MS from the Norwegian MS registry.
Information about the MS disease at 5 years after randomization | 5 years after randomization
  Disability status assessed with the Extended Disability Status Scale from the Norwegian MS registry, information about previous and current treatment for MS, previous attack phases, first diagnosis of MS from the Norwegian MS registry.
Excessive daytime sleepiness at baseline | Baseline
  Assessed with the Epworth Sleepiness Scale, a eight item questionnaire. The eight items represent real-life situations where the participants must rate their chance of dozing off using a 4-point scale from 0 to 3. Higher scores indicate higher chance of dozing off. Total score indicates the extent of self-reported sleep propensity.
Subjective cognitive disfunction at baseline | Baseline
  Assessed with the Cognitive Complaints in Bipolar Disorder Rating Assessment (COBRA), a 16-item self-reported instrument of subjective cognitive dysfunctions including executive function, processing speed, working memory, verbal learning and memory, attention/concentration and mental tracking. Items are rated using a 4-point scale. The higher the score, the more subjective complaints. Although the assessment was initially introduced for use with individuals with bipolar disorders, the rating can be used in other clinical populations
Subjective executive functions at baseline | Baseline
  Assessed with the Behavior Rating Inventory of Executive Function for Adults, a 75 item questionnaire that that captures views of an adult's executive functions or self-regulation in his or her everyday environment. Items are rated on a 3-point scale (Never a problem - sometimes a problem - often a problem).
Subjective executive functions at 9 weeks after randomization | 9 weeks after randomization
  Assessed with the Behavior Rating Inventory of Executive Function for Adults, a 75 item questionnaire that that captures views of an adult's executive functions or self-regulation in his or her everyday environment. Items are rated on a 3-point scale (Never a problem - sometimes a problem - often a problem).
Subjective executive functions at 33 weeks after randomization | 33 weeks after randomization
  Assessed with the Behavior Rating Inventory of Executive Function for Adults, a 75 item questionnaire that that captures views of an adult's executive functions or self-regulation in his or her everyday environment. Items are rated on a 3-point scale (Never a problem - sometimes a problem - often a problem).
Subjective executive functions at 61 weeks after randomization | 61 weeks after randomization
  Assessed with the Behavior Rating Inventory of Executive Function for Adults, a 75 item questionnaire that that captures views of an adult's executive functions or self-regulation in his or her everyday environment. Items are rated on a 3-point scale (Never a problem - sometimes a problem - often a problem).
Subjective disability status at baseline | Baseline
  Assessed with the Patient-Determined Disease Steps (PDDS), a questionnaire where the participants are asked to choose one out of nine alternatives that bests describes their current disability status
Fatigue before and after cognitive testing at baseline | Baseline
  Feelings of state fatigue assessed with a single question (i.e "How much fatigue do you feel right now"). The participants are asked to rate their feelings of fatigue on a 4-point scale from 0=no fatigue, to 4=severe fatigue right before cognitive testing and immediately after cognitive testing.
Fatigue before and after cognitive testing at 9 weeks | 9 weeks after randomization
  Feelings of state fatigue assessed with a single question (i.e "How much fatigue do you feel right now"). The participants are asked to rate their feelings of fatigue on a 4-point scale from 0=no fatigue, to 4=severe fatigue right before cognitive testing and immediately after cognitive testing.
Fatigue before and after cognitive testing at 33 weeks | 33 weeks after randomization
  Feelings of state fatigue assessed with a single question (i.e "How much fatigue do you feel right now"). The participants are asked to rate their feelings of fatigue on a 4-point scale from 0=no fatigue, to 4=severe fatigue right before cognitive testing and immediately after cognitive testing.
Fatigue before and after cognitive testing at 61 weeks | 61 weeks after randomization
  Feelings of state fatigue assessed with a single question (i.e "How much fatigue do you feel right now"). The participants are asked to rate their feelings of fatigue on a 4-point scale from 0=no fatigue, to 4=severe fatigue right before cognitive testing and immediately after cognitive testing.
Perceived performance after cognitive testing at baseline | Baseline
  Perceived performance after cognitive testing will be assessed with a single question (i.e. How did you feel like you performed on the test?) rated on a 10-point scale (1=very bad, 10=very good performance)
Perceived performance after cognitive testing at 9 weeks | 9 weeks after randomization
  Perceived performance after cognitive testing will be assessed with a single question (i.e. How did you feel like you performed on the test?) rated on a 10-point scale (1=very bad, 10=very good performance)
Perceived performance after cognitive testing at 33 weeks | 33 weeks after randomization
  Perceived performance after cognitive testing will be assessed with a single question (i.e. How did you feel like you performed on the test?) rated on a 10-point scale (1=very bad, 10=very good performance)
Perceived performance after cognitive testing at 61 weeks | 61 weeks after randomization
  Perceived performance after cognitive testing will be assessed with a single question (i.e. How did you feel like you performed on the test?) rated on a 10-point scale (1=very bad, 10=very good performance)
Perceived exertion after cognitive testing at baseline | Baseline
  Perceived exertion after cognitive testing will be assessed with a single question (i.e. How much exertion did you feel during the test?) rated on a 10-point scale (1=no exertion at all, 10=very much exertion)
Perceived exertion after cognitive testing at 9 weeks | 9 weeks after randomization
  Perceived exertion after cognitive testing will be assessed with a single question (i.e. How much exertion did you feel during the test?) rated on a 10-point scale (1=no exertion at all, 10=very much exertion)
Perceived exertion after cognitive testing at 33 weeks | 33 weeks after randomization
  Perceived exertion after cognitive testing will be assessed with a single question (i.e. How much exertion did you feel during the test?) rated on a 10-point scale (1=no exertion at all, 10=very much exertion)
Perceived exertion after cognitive testing at 61 weeks | 61 weeks after randomization
  Perceived exertion after cognitive testing will be assessed with a single question (i.e. How much exertion did you feel during the test?) rated on a 10-point scale (1=no exertion at all, 10=very much exertion)
Insomnia symptoms and severity at baseline | Baseline
  Assessed with the Bergen Insomnia Scale (BIS). BIS comprises six items that assesses symptoms of insomnia based on the insomnia criteria found in the Diagnostic and Statistical Manual of Mental Disorders-IVTR (American Psychiatric Association).
Insomnia symptoms and severity at 9 weeks | 9 weeks after randomization
  Assessed with the Bergen Insomnia Scale (BIS). BIS comprises six items that assesses symptoms of insomnia based on the insomnia criteria found in the Diagnostic and Statistical Manual of Mental Disorders-IVTR (American Psychiatric Association).
Insomnia symptoms and severity at 33 weeks | 33 weeks after randomization
  Assessed with the Bergen Insomnia Scale (BIS). BIS comprises six items that assesses symptoms of insomnia based on the insomnia criteria found in the Diagnostic and Statistical Manual of Mental Disorders-IVTR (American Psychiatric Association).
Insomnia symptoms and severity at 61 weeks | 61 weeks after randomization
  Assessed with the Bergen Insomnia Scale (BIS). BIS comprises six items that assesses symptoms of insomnia based on the insomnia criteria found in the Diagnostic and Statistical Manual of Mental Disorders-IVTR (American Psychiatric Association).
Pain map with numeric rating scale at baseline | Baseline
  Presence of pain beyond everyday mundane pain, that have lasted longer than 3 months will be assessed with a single yes/no question. Location of pain will be assessed with a pain map, and levels of pain will be assessed with a 11-point numeric rating scale (0 = no pain to 10= severe pain.)
Frequency of alcohol use at baseline | Baseline
  Assessed with the Alcohol Use Disorders Identification Test - Consumption (AUDIT-C), a three-item self-report questionnaire assessing frequency of alcohol use (0=never, 4=four times each week or more), number of units typical for a drinking day (0=1-2 units, 4=10 or more units), and frequency of binge-drinking (0=never, 4=daily or almost daily). It is a short-version of the 10-item AUDIT developed by the World Health Organization
Frequency of alcohol use at 9 weeks | 9 weeks after randomization
  Assessed with the Alcohol Use Disorders Identification Test - Consumption (AUDIT-C), a three-item self-report questionnaire assessing frequency of alcohol use (0=never, 4=four times each week or more), number of units typical for a drinking day (0=1-2 units, 4=10 or more units), and frequency of binge-drinking (0=never, 4=daily or almost daily). It is a short-version of the 10-item AUDIT developed by the World Health Organization
Frequency of alcohol use at 33 weeks | 33 weeks after randomization
  Assessed with the Alcohol Use Disorders Identification Test - Consumption (AUDIT-C), a three-item self-report questionnaire assessing frequency of alcohol use (0=never, 4=four times each week or more), number of units typical for a drinking day (0=1-2 units, 4=10 or more units), and frequency of binge-drinking (0=never, 4=daily or almost daily). It is a short-version of the 10-item AUDIT developed by the World Health Organization
Frequency of alcohol use at 61 weeks | 61 weeks after randomization
  Assessed with the Alcohol Use Disorders Identification Test - Consumption (AUDIT-C), a three-item self-report questionnaire assessing frequency of alcohol use (0=never, 4=four times each week or more), number of units typical for a drinking day (0=1-2 units, 4=10 or more units), and frequency of binge-drinking (0=never, 4=daily or almost daily). It is a short-version of the 10-item AUDIT developed by the World Health Organization
Self reported quality of life at baseline | Baseline
  Assessed with the 12-Item Short Form Survey (SF-12). SF-12 The SF-12 is a self-reported outcome measure assessing the impact of health on an individual's everyday life, and is a measure of quality of life. The SF-12 is a shortened version of the SF-36.
Self reported quality of life at 9 weeks | 9 weeks after randomization
  Assessed with the 12-Item Short Form Survey (SF-12). SF-12 The SF-12 is a self-reported outcome measure assessing the impact of health on an individual's everyday life, and is a measure of quality of life. The SF-12 is a shortened version of the SF-36.
Self reported quality of life at 33 weeks | 33 weeks after randomization
  Assessed with the 12-Item Short Form Survey (SF-12). SF-12 The SF-12 is a self-reported outcome measure assessing the impact of health on an individual's everyday life, and is a measure of quality of life. The SF-12 is a shortened version of the SF-36.
Self reported quality of life at 61 weeks after randomization | 61 weeks after randomization
  Assessed with the 12-Item Short Form Survey (SF-12). SF-12 The SF-12 is a self-reported outcome measure assessing the impact of health on an individual's everyday life, and is a measure of quality of life. The SF-12 is a shortened version of the SF-36.
General health state at baseline | Baseline
  Assessed with Euroqol-5D, a 5-item self-report questionnaire for general health state on a 0 to 5 likert scale. It measures levels of problems with walking, performing self-care, doing usual activities, pain/discomfort, and anxiety/depression. It is widely used across Europe in assessments of health resources utilization as it allows measurement of Quality Adjusted Life Years (QALYs) in individuals presenting with a wide range of physical and mental disorders
General health state at 9 weeks | 9 weeks after randomization
  Assessed with Euroqol-5D, a 5-item self-report questionnaire for general health state on a 0 to 5 likert scale. It measures levels of problems with walking, performing self-care, doing usual activities, pain/discomfort, and anxiety/depression. It is widely used across Europe in assessments of health resources utilization as it allows measurement of Quality Adjusted Life Years (QALYs) in individuals presenting with a wide range of physical and mental disorders
General health state at 33 weeks | 33 weeks after randomization
  Assessed with Euroqol-5D, a 5-item self-report questionnaire for general health state on a 0 to 5 likert scale. It measures levels of problems with walking, performing self-care, doing usual activities, pain/discomfort, and anxiety/depression. It is widely used across Europe in assessments of health resources utilization as it allows measurement of Quality Adjusted Life Years (QALYs) in individuals presenting with a wide range of physical and mental disorders
General health state at 61 weeks | 61 weeks after randomization
  Assessed with Euroqol-5D, a 5-item self-report questionnaire for general health state on a 0 to 5 likert scale. It measures levels of problems with walking, performing self-care, doing usual activities, pain/discomfort, and anxiety/depression. It is widely used across Europe in assessments of health resources utilization as it allows measurement of Quality Adjusted Life Years (QALYs) in individuals presenting with a wide range of physical and mental disorders
Opinion on negative effects of the intervention at 9 weeks | 9 weeks after randomization
  Assessed with the Negative Effects Questionnaire (NEQ), a self-report measure that contains 20 items that are scored on a five-point Likert-scale (rated 0-4) where higher scores indicate higher levels of negative effects. After each item, the individual is asked whether they consider the effect to be caused by the intervention received or caused by other circumstances (yes/no), as well as one open-ended question
Opinion on negative effects of the intervention at 61 weeks | 61 weeks after randomization
  Assessed with the Negative Effects Questionnaire (NEQ), a self-report measure that contains 20 items that are scored on a five-point Likert-scale (rated 0-4) where higher scores indicate higher levels of negative effects. After each item, the individual is asked whether they consider the effect to be caused by the intervention received or caused by other circumstances (yes/no), as well as one open-ended question
Use of therapeutic techniques at 33 weeks | 33 weeks after randomization
  Assessed with the Use of Sleep Strategies (USS), a six item self-report questionnaire developed to measure how often individuals use six different therapeutic techniques (keep a stable rise time, refrain from sleeping during daytime, use the bed and bedroom only for sleeping, practiced sleep restriction, practiced stimulus control) and their perception of its utility. The techniques are integral to CBT-I but are also described in sleep psychoeducation or hygiene programmes
Use of therapeutic techniques at 61 weeks | 61 weeks after randomization
  Assessed with the Use of Sleep Strategies (USS), a six item self-report questionnaire developed to measure how often individuals use six different therapeutic techniques (keep a stable rise time, refrain from sleeping during daytime, use the bed and bedroom only for sleeping, practiced sleep restriction, practiced stimulus control) and their perception of its utility. The techniques are integral to CBT-I but are also described in sleep psychoeducation or hygiene programmes
Self-reported medication usage at baseline | Baseline
  Dose, timing, and type of prescribed and unsubscribed medications
Self-reported previous and current physical and mental disorders at baseline | Baseline
  Assessed by checking of a list of 20 common medical conditions, and 9 common mental disorders
Self-reported physical activity at baseline | Baseline
  Number of physical activities per week at moderate and/or strenuous intensity, and duration of the activities
Self-reported Body Mass Index (BMI) at baseline | Baseline
  One question assessing height and one question assessing weight
Self-reported internet and media usage at baseline | Baseline
  Familiarity with use of the internet at baseline and electronic media use (five items) over time. These ratings will be used in subsidiary analyses as for example, how baseline skills in using the internet may affect engagement with internet interventions.
Self-reported previous treatments for mental disorders at baseline | Baseline
  Number of previous treatments, number of prescribed medications for mental disorders
Self-reported previous treatments for insomnia at baseline | Baseline
  Number of previous treatments, number of prescribed medications for insomnia
Self-reported duration of sleep problems at baseline | Baseline
  One item assessing for how long the current sleep problem have lasted in years and months

CONTACTS AND LOCATIONS:
Overall Officials: Håvard Kallestad, PhD, Principal Investigator — Senior clinical psychologist and researcher
Locations (1):
- St.Olavs Hospital, Trondheim, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Saksvik SB, Ronhovde LM, Ytrehus-Lynum K, Langsrud K, Olsen A, das Nair R, Lydersen S, Holthe JG, Halvorsen JO, Morken G, Ritterband LM, Bo L, Kallestad H. Digital cognitive behavioral therapy for insomnia compared with digital patient education about insomnia in people with multiple sclerosis in Norway: study protocol for a randomized controlled trial. Sleep Adv. 2025 Oct 31;6(4):zpaf075. doi: 10.1093/sleepadvances/zpaf075. eCollection 2025. PMID 41278218